CLINICAL TRIAL: NCT06333119
Title: The Relationship Between Urinary Incontinence and Motor Symptoms in Individuals With Stroke
Brief Title: The Relationship Between Urinary Incontinence and Motor Symptoms
Status: Completed | Type: Observational
Sponsor: Pinar Yasar (Other)
Responsible Party: Sponsor-Investigator, Pinar Yasar, Research assistant, Physiotherapist, Suleyman Demirel University
Organization: Suleyman Demirel University (Other)
Other Study IDs: 72867572-050.01.04-320
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Stroke; Urinary Incontinence; Motor Skills Disorders
Keywords: stroke; urinary incontinence; spasticity; balance; gait
MeSH Terms: conditions — Stroke; Urinary Incontinence; Motor Skills Disorders; Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- individuals with stroke
  Interventions: Diagnostic Test: modified rankin scale

INTERVENTIONS:
Diagnostic Test: modified rankin scale — Modified Rankin Scale: The functional status of individuals with stroke is determined by this scale.
  Modified Ashworth Scale: It allows determining the severity of spasticity. Tinetti Balance and Gait Scale: This scale helps determine the risk of falling by evaluating balance and gait.
  Danish Prostatic Symptom Score: It allows to evaluate the storage and urinary functions of the bladder.
  Other Names: modified ashworth scale; Tinetti Balance and Gait Scale; Danish Prostatic Symptom Score

SUMMARY:
There is no study in the literature examining the relationship between urinary incontinence and motor symptoms in individuals with stroke. The aim of this study is to determine the relationship between urinary incontinence and spasticity, balance and walking, which negatively affect quality of life and functional performance after stroke.

DETAILED DESCRIPTION:
Evaluation parameters used in the study:

Modified Rankin Score 24 hours pad test Tinetti Balance and Gait Scale Modified Ashworth scale Danish Prostatic Symptom Score

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years old, having a stroke history of at least 3 months, having had only one stroke, scoring between 0-2 points according to MRS, being able to stand and walk independently or with a walking aid, being able to speak Turkish.

Exclusion Criteria:

* Those with incomprehensible speech disorders,
* Those who have additional neurological diseases other than stroke,
* orthopedic, cardiovascular, etc., which may cause balance disorders. those with illnesses,
* those who are pregnant,
* Those with vision and hearing loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: individuals with stroke
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
relationship with between urinary incontinence and motor symptoms | 4 months
  correlation analysis was done.

CONTACTS AND LOCATIONS:
Overall Officials: Pinar Yasar, Study Director — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It was decided not to share the data, taking into account the personal data protection law.